CLINICAL TRIAL: NCT04774133
Title: Radioinduced Modifications of Lymphocyte Subpopulations Involved in Resistence and Escape Mechanisms to Radiation Therapy of Localized Prostate Cancer.
Brief Title: The Immunodynamic Effect of Radiotherapy in Prostate Cancer Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: Paola Nisticò (Unknown); Iole Cordone (Unknown); Adriana Faiella (Unknown); Paola Trono (Unknown); Serena Masi (Unknown); Roberta Merola (Unknown); Anna Antenucci (Unknown); Maria Laura Foddai (Unknown); Maria Consiglia Ferriero (Unknown); Diana Giannarelli (Unknown); Paolo Di Ridolfi (Unknown)
Responsible Party: Principal Investigator, Giuseppe Sanguineti, Radioinduced Modifications of Lymphocyte Subpopulations Involved in Resistence and Escape Mechanisms to Radiation Therapy of Localized Prostate Cancer., Regina Elena Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1163/18
Record Dates: First submitted 2021-02-23; First posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Prostatic Neoplasm
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Blood sample — Pazients will undergo to blood samples at predefined times

SUMMARY:
Radiotherapy has an important role in the treatment of prostate cancer both as curative treatment and postoperative or salvage ones. Several studies demonstrated a significant reduction of lymphocytes during RT but there are only a few studies monitoring these cells in the treatment of prostate cancer. This study will enroll 50 patients with hystologically proven prostate cancer who will undergo to radiotherapy according to Institutional protocols.

This study aims to evaluate the effect of RT on immuno-regulatory B, NK, T, B and T lymphocyte subpopulations (Breg and Treg) and plasma cells, quantitative / qualitative changes,their correlations with the clinical course of the disease and acute and late toxicity. In parallel, using multicolor panels (12 colors) we will evaluate the expression of inhibitory checkpoints and TGFβ signaling.

The final objective is to identify new therapeutic targets to be combined with RT.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented prostatic cancer
* Indication to perform radiotherapy treatment
* Age over 18 years
* Informed consent

Exclusion Criteria:

* Hematological diseases
* Autoimmune diseases
* Previous neoplasias
* Prior chemotherapy or other therapies that may have violated the hematopoietic organs
* Patient's refusal to undergo periodic blood samples

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-02-14 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
to quantify the variation in lymphocyte subpopulations T, NK, B, Breg and Treg, | 12 months
  quantitative variation

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Sanguineti, Principal Investigator — IFO
Locations (1):
- IRCSS Regina Elena, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided